CLINICAL TRIAL: NCT00832923
Title: Improving Asthma Care Through Parental Empowerment: Effect on Healthcare Utilization and Parent Self-Efficacy
Brief Title: Improving Asthma Care Through Parental Empowerment
Acronym: PEPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Stephen J. Teach, MD, MPH, Chief, Division of Allergy and Immunology, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RAC #207
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Asthma
Keywords: parental empowerment; parent self-efficacy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine IMPACT DC care (No Intervention): Participants receive standard asthma education as routine for IMPACT DC
- Enhanced care PEPAC Intervention (Experimental)
  Interventions: Behavioral: PEPAC

INTERVENTIONS:
Behavioral: PEPAC — The proposed enhancement of the IMPACT DC intervention will consist of three key components: (1) an enhanced IMPACT DC Asthma Clinic visit; (2) short-term case management to increase the rate of primary care follow-up visits in the first month after the IMPACT DC Asthma Clinic visit; and (3) training in an "asthma care toolkit" to improve communication around asthma care with the child's primary care provider.
  Arms: Enhanced care PEPAC Intervention

SUMMARY:
The overall aim of this study will be to perform a prospective randomized clinical trial of an enhanced version of the IMPACT DC intervention involving short-term case management to facilitate PCP follow-up appointments and to provide education for parents about how to communicate more effectively with their children's PCPs as a means (1) to improve the rate of utilization of primary care services for ongoing asthma care and (2) to enhance the self-efficacy of parents in their interactions with their children's provider regarding the child's asthma care needs in 150 parents of high risk children referred within the IMPACT DC Asthma Clinic.

DETAILED DESCRIPTION:
Asthma is the most common chronic disease of childhood, and it disproportionately affects urban, minority, and disadvantaged children. When implemented correctly, existing evidence-based guidelines from the National Heart, Lung, and Blood Institute (NHLBI) improve pediatric asthma care and outcomes. One key component of these guidelines is the importance of longitudinal care as part of a partnership among patient, parents, and a healthcare provider. Such a partnership depends on effective communication of healthcare status by parents to providers. Improving the communication skills of inner-city parents may improve their ability to obtain more effective longitudinal asthma care within their primary care homes and thereby to improve their child's asthma health outcomes. IMPACT DC ("Improving Pediatric Asthma Care in the District of Columbia") is a locally validated emergency department (ED) based intervention that improves multiple measures of asthma care and outcomes through an intensive short-term program of asthma education, medical care, and care coordination. In spite of these successes, achieving increased subsequent contact and partnership with primary care providers (PCPs) for asthma care after the intervention has not been successful. Therefore, for the current study, we propose to assess the effectiveness of an enhanced version of the existing IMPACT DC intervention consisting of short-term case management by trained asthma educators.

ELIGIBILITY:
Inclusion Criteria:

* ages between 12 months and 12 years, inclusive
* prior physician diagnosed asthma
* ability of the parent to identify a specific PCP for their child
* public insurance covering the child
* parent/guardian available for interview

Exclusion Criteria:

* significant medical co-morbidities
* enrollment in another asthma research intervention study
* unavailability for telephone follow-up
* primary language of the caregiver other than English

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Utilization of Primary Care Provider | 2 months & 6 months after visit

SECONDARY OUTCOMES:
Parental Self-efficacy in communicating about Asthma care with child's primary care provider | 2 months & 6 months after visit

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Research Institute, Washington D.C., District of Columbia, United States